CLINICAL TRIAL: NCT03006770
Title: Efficacy, Tolerability and Safety of Intramuscular Injections of PLX PAD for the Treatment of Subjects With Critical Limb Ischemia (CLI) With Minor Tissue Loss Who Are Unsuitable for Revascularization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pluristem Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLX-CLI-03
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Critical Limb Ischemia (CLI)
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PLX-PAD (Experimental): PLX-PAD will be administered via 30 IM injections (0.5 mL each). Each subject will be treated twice, with an interval of 8 weeks between treatments.
  Interventions: Biological: PLX-PAD
- Placebo (Placebo Comparator): Placebo will be administered via 30 IM injections (0.5 mL each). Each subject will be treated twice, with an interval of 8 weeks between treatments.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PLX-PAD — Local intramuscular (IM) injections of PLX-PAD in the index leg.
  Arms: PLX-PAD
Biological: Placebo — Local intramuscular (IM) injections of Placebo in the index leg.
  Arms: Placebo

SUMMARY:
This will be a randomized, placebo-controlled, parallel group, multicenter, Phase III study.The study aims to evaluate the Efficacy, Tolerability and Safety of Intramuscular Injections of PLX PAD for the Treatment of Subjects with Critical Limb Ischemia (CLI) with Minor Tissue Loss (Rutherford Category 5) who are Unsuitable for Revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female subjects between ages 45-99 years of age.
2. CLI, with minor tissue loss up to the ankle level (Rutherford Category 5)
3. Ankle pressure (AP) ≤70 mmHg or TP ≤50 mmHg in the index leg. (If a subject has ABI >1.4 and TP is not measureable, inclusion may be based on TcPO2 ≤30 mmHg)
4. Subject unsuitable for revascularization (by any method) in the index leg.
5. Ischemic lesions in the index leg stable for at least 2 weeks.
6. Ischemic ulcers in the index leg without tendon or bone exposure (unless secondary to a minor amputation).
7. Under treatment for cardiovascular risk factors: hypertension, hyperlipidemia, diabetes, in accordance with applicable guidelines. Concomitant therapy with a statin and an anti-platelet agent for at least 2 weeks prior to randomization.
8. Women of childbearing potential must have a negative serum pregnancy test at screening and must be willing to use at least one highly effective birth control method throughout the study.
9. Subject understood, agreed and provided informed consent. Patients must give written informed consent before any assessment is performed .

Exclusion Criteria:

1. Non-atherosclerotic PAD (e.g. Buerger's disease).
2. CLI with major tissue loss (Rutherford Category 6) in either leg.
3. Evidence of active infection (e.g., cellulitis, osteomyelitis).
4. Subject having undergone surgical revascularization or major amputation less than 1 month prior to screening, or endovascular revascularization or minor amputation less than 2 weeks prior to screening.
5. Planned or potential need for major/minor amputation or any revascularization within 1 month of study entry upon investigator's judgment.
6. Aorto-iliac stenosis or common femoral artery stenosis ≥70%, or otherwise suspicion of inadequate inflow to the leg.
7. Life expectancy of less than 6 months.
8. Stroke or acute myocardial infarction/unstable angina within 3 months prior to screening.
9. Severe congestive heart failure symptoms (New York Heart Association [NYHA] class III-IV).
10. Uncontrolled severe hypertension.
11. Diabetes mellitus with HbA1c >10%.
12. Current or history of proliferative retinopathy.
13. Known Hepatitis B virus or Hepatitis C virus or acquired immunodeficiency syndrome (AIDS) infections.
14. Subjects with international normalized ratio (INR) >2.
15. Subject on renal replacement therapy or planned to start renal replacement therapy within 3 months of first screening visit.
16. Subject is currently enrolled in, or has not yet completed a period of at least 30 days since ending another investigational device or drug trial(s), unless in long-term follow-up phase.
17. Use of hyperbaric oxygen therapy, prostanoids, spinal cord stimulation, lumbar sympathectomy, wound dressing containing cells or growth factors, or topical platelet derived growth factor.
18. Known allergies to any of the following: DMSO, human serum albumin, bovine serum albumin.
19. History of allergic/hypersensitivity reaction to any substance having required hospitalization and/or treatment with IV steroids/epinephrine.
20. Pulmonary disease requiring supplemental oxygen treatment on a daily basis.
21. Active malignancy or history of malignancy within 5 years prior to study entry.
22. In the opinion of the investigator, the subject is unsuitable for participating in the study.
23. Chronic liver disease Child Pugh class B\C

Ages: 45 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Time to major amputation or death (AFS) | Up to 36 months from enrollment

SECONDARY OUTCOMES:
Time to first occurrence of any of the events (in index leg)-major amputation, revascularization due to worsening of CLI, All-cause mortality. | Up to 36 months from enrollment
Time to major amputation of the index leg. | Up to 36 months from enrollment
Change from baseline in ischemic pain as assessed by numerical rating scale (NRS) at 6 months. | 6 months from enrollment
  NRS measures the intensity or magnitude of sensations and subject feelings and the relative strength of attitudes and opinions about specific stimuli, on a scale of 0 to 10 with a score of zero denoting "no pain at all" and a score of 10 denoting "worst possible pain".
Proportion of subjects with complete healing of all ischemic lesions i.e., ulcers and necroses in the index leg at 12 months. | 12 months from enrollment
Time (days) from randomization to occurrence of death. | Up to 36 months from enrollment

CONTACTS AND LOCATIONS:
Locations (57):
- United States (14):
  - UCI Medical Center 101 The City Drive S. Bldg 55 Rm 334 Orange, CA 92868, Irvine, California
  - Cedars Sinai Medical Center,LA,Beverly Hills,8536 Wilshire Boulevard, Third Floor, Los Angeles, California
  - Vascular Center ∣ Department of Surgery ∣ UC Davis Health 4860 Y street, Sacramento, CA suite #3400, 95817, Sacramento, California
  - Vascular Center,Department of Surgery,UC Davis Health,4860 Y street, Sacramento, California
  - University of Miami Leonard M.Miller School of Medicine (UMMSM)-UHealth Pulmonary and Critical Care Medicine-Rosenstiel Building Location, Miami, Florida
  - Miami Cardiac and Vascular Institute Baptist Health South Florida, Miami, Florida
  - Tufts Medical Center (TMC) (Tufts-New England Medical Center), Boston, Massachusetts
  - Room S3-746, Dept of Surgery, UMASS Medical School, 55 Lake Ave North., Worcester, Massachusetts
  - Holy Medical Center, Teaneck, New Jersey
  - Northwell Health Comprehensive Wound Healing Center, Lake Success, New York
  - Mount Sinai St. Luke's hospital, New York, New York
  - Duke University Medical Center,Durham,2424 Erwin Road Hock Plaza, Durham, North Carolina
  - Austin Heart Clinical Research, Austin, Texas
  - Department of Plastic Surgery ,Ut Southwestern Medical Center, Dallas, Texas
- Bulgaria (8):
  - UMHAT "Virgin Mary" EOOD,Clinic of Vascular Surgery, Burgas
  - MHAT Sveti Nokolay Chudotvorets EOOD - Lom,Surgery Department,Address 2, Todor Kableshkov str., Lom
  - UMHAT "St. Georgi" EAD,Clinic: Vascular Surgery and Angiology 66 "Peshtersko Shosse" Blvd., 8th floor, Hirurgicheski blok, Plovdiv
  - UMBAL Kanev AD - Ruse,Department of Vascular Surgery Address: 2, Nezavisimost str, Rousse
  - UMHAT "Medica" Ruse Department of Vascular Surgery 35, "Riga", Str Post code: 7013 Ruse, Bulgaria, Rousse
  - MHAT National Heart Hospital EAD,Clinic of Vascular Surgery and angiology, Sofia
  - Acibadem City Clinic MHAT Tokuda, Vascular Surgery and Angiology 51B "Nikola Vaptzarov" Blvd, Sofia
  - UMHAT "St. Ekaterina" EAD, Departement of Vascular Surgery, Sofia
- Czechia (5):
  - Cevni ambulance, Hodonín
  - Angiologicka ambulance, Ostrava Dubina
  - Vseobecna Fakultni Nemocnice v Praze, Prague
  - Intitute of Clinical and Experimental Medicine, Prague
  - Krajska zdravotni a.s., Masarykova nemocnice o.z., Ústí nad Labem
- Germany (10):
  - Klinik und Poliklinik für Angiologie Universitätsklinikum Leipzig AöR Liebigstr. 20 04103 Leipzig, Germany, Leipzig, Saxony
  - Medinos Klinikum Sonneberg Abteilung für Kardiologie/Angiologie - Studienambulanz Neustadter Straße 61 96515 Sonneberg Germany, Sonneberg, Thuringia
  - Universitats-Herzzentrum Freiburg, Bad Krozingen
  - Charite Centrum fur Herz - Kreislauf - und Gefassmedizin - Campus Benjamin Franklin, Berlin
  - HELIOS Klinikum Berlin-Buch, Klinik fur Angiologie, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Heinrich-Heine-Universitaet Duesseldorf - Universitaetsklinikum Duesseldorf (UKD), Düsseldorf
  - Asklepios Klinik St.Georg-Angiologische Ambulanz, Hamburg
  - Klinik Kösching Krankenhausstr. 19, 85092 Kösching Germany, Kösching
  - Universitaetsklinikum Muenster, Münster
- Hungary (6):
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár, Fejér
  - Szent Imre Egyetemi Oktato Korhaz, Budapest
  - Flor Ferenc County Hospital, Kistarcsa
  - B-A-Z County and University Teaching Hospital, Miskolc
  - Josa Andras Megyei Korhaz, Nyíregyháza
  - Pecsi Tudomanyegyetem (PTE) Altalanos Orvostudomanyi Kar (AOK) (University of Pecs Medical School), Pécs
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Blood Vessel Day Care at Clalit Community Horev Center, Horev Center, Haifa
  - Vascular Surgery Department, Hadassah Ein Karem MC, Jerusalem
  - Vascular Surgery Department Rabin Medical Center Beilinson Hospital, 39 Jabotinski St. Petah Tikva Israel 4941492, Petah Tikva
  - The Cardiological Department, The Baruch Padeh Medical Center, Poria Illit
- North Macedonia (3):
  - Acibadem Sistina Hospital,Thoracic and Vascular Surgery, Skopje
  - Re-Medika General Hospital,Cardiovascular Surgery, Skopje
  - Special Hospital for Surgical Diseases Zan Mitrev Clinic ,Cardiovascular Surgery, Skopje
- Poland (2):
  - Cathedra and Clinic of Vascular Surgery and Angiology-Klinika Chirurgii Naczyniowej i Angiologii, Lublin
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Osrodek Badawczo-Rozwojowy,Intensywnego Nadzoru Kardlologleznego,, Wroclaw
- United Kingdom (4):
  - Vascular Research Clinical Research Centre Beaufort Way Southmead Hospital Westbury on Trym Bristol, Bristol
  - Hull And East Yorkshire Women And Children's Hospital-Hull And East Yorkshire Hospitals Nhs Trust, Hull
  - Kings College Hospital, London
  - Department of Vascular Research, St George's Hospital, London

REFERENCES:
- [Derived] Norgren L, Weiss N, Nikol S, Lantis JC, Patel MR, Hinchliffe RJ, Reinecke H, Volk HD, Reinke P, Fadini GP, Ofir R, Rothenstein D, Halevy N, Karagjozov M, Rundback JH. PACE: randomized, controlled, multicentre, multinational, phase III study of PLX-PAD for critical limb ischaemia in patients unsuitable for revascularization: randomized clinical trial. Br J Surg. 2024 Jan 31;111(2):znad437. doi: 10.1093/bjs/znad437. PMID 38294084
- [Derived] Norgren L, Weiss N, Nikol S, Hinchliffe RJ, Lantis JC, Patel MR, Reinecke H, Ofir R, Rosen Y, Peres D, Aberman Z. PLX-PAD Cell Treatment of Critical Limb Ischaemia: Rationale and Design of the PACE Trial. Eur J Vasc Endovasc Surg. 2019 Apr;57(4):538-545. doi: 10.1016/j.ejvs.2018.11.008. Epub 2019 Jan 25. PMID 30686676